CLINICAL TRIAL: NCT04851743
Title: Effects on Neuromuscular Function After Dry Needling in Myofascial Trigger Points in the Gastrocnemius Muscles: A Randomized Within-Participant Clinical Trial
Brief Title: Effects on Neuromuscular Function After Dry Needling in Myofascial Trigger Points in the Gastrocnemius Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Director Human Anatomy Laboratory, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBAS-2018-11B
Record Dates: First submitted 2020-09-28; First posted 2021-04-20 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2020-09

CONDITIONS: Myofascial Trigger Point Pain
Keywords: dry needling; gastrocnemius; myofascial trigger point
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: A randomized within-participant clinical trial
Who Masked: Outcomes Assessor
Masking Description: the assessor will not know if patients have received the dry needling technique or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling Group (Experimental): Participants will be used as their own controls, with 1 lower extremity randomly receiving intervention. The experimental extremity will received a single treatment session of TrP dry needling as follows: the therapist will located the TrP and will applied manual compression until the participant will reported pain. After that, dry needling technique will be performed on the TrPs for 60 seconds.
  Interventions: Other: Dry needling
- Control Group (No Intervention): Participants will be used as their own controls, with 1lower extremity randomly receiving intervention. The control extremity did not receive any intervention, and outcomes were assessed 2 minutes apart.

INTERVENTIONS:
Other: Dry needling — The experimental extremity will received a single treatment session of TrP dry needling as follows: the therapist will located the TrP and will applied manual compression until the participant will reported pain. After that, dry needling technique will be performed on the TrPs for 60 seconds.
  Arms: Dry needling Group

SUMMARY:
Trigger points (TrPs) are a common musculoskeletal cause of local and referred muscle pain, as well as local inflammation in the muscle and fascia. From a clinical and sensory viewpoint, TrPs may be classified as active or latent. The principal difference is the reproduction of symptoms experienced by an individual (active) with or without stimulation. Local and referred pain elicited from latent TrPs may be transient in duration upon stimulation, and latent TrPs may be present without spontaneous symptoms.

Both active and latent TrPs induce motor dysfunctions such as stiffness, restricted range of motion, and accelerated fatigability in the affected muscle. The interrater reliability of manual identification of latent TrPs in the calf muscles has been found to range from small to moderate. The clinical relevance of latent TrPs has increased in the last decade,4 and some studies have investigated the effects of treating them. Among all manual therapies targeted to latent TrPs, ischemic compression, or TrP pressure release, is the most commonly used. Although TrPs may affect any muscle, the gastrocnemius muscle may be the most susceptible in the lower extremity to developing them. It has been reported that 13% to 30% of the asymptomatic population has latent TrPs in these muscles, and their presence may affect sport practice.

The purpose of this study will be to evaluate changes in neuromuscular function, pain perception, and basic physical properties in myofascial trigger points (TrPs) after a single treatment session of dry needling in the gastrocnemius muscle.

A randomized within-participant clinical trial with a blinded assessor will be conducted. 50 asymptomatic volunteers (100 gastrocnemius-muscle) with MrPs gastrocnemius-muscle TrPs will bilaterally explored. Each extremity will be randomly assigned to the control group (no treatment) or the experimental group (60 seconds of dry needling over each TrP). Neuromuscular function of the gastrocnemius muscle will be assessed using a MyotonPro and a tensiomyography. Muscle flexibility will be analyzed using the lunge test and the passive ankle range of motion. The strength will be determined with a handheld dynamometer (MicroFET2). Pain perception will be analyzed with a 0-to-10 numerical pain rating scale and determination of pressure pain thresholds over each latent TrP.

ELIGIBILITY:
Inclusion Criteria:

* A TrP will be diagnosed using the following criteria: palpable taut band, presence of a painful spot in the taut band, and referred pain on palpation of the spot.

Exclusion Criteria:

* Participants were excluded if they reported any pain symptoms in the lower extremities in the previous year.
* They were also excluded if they presented previous surgical interventions, previous lower-extremity injury, any underlying medical disease, pregnancy, or muscle soreness after vigorous exercise.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Neuromuscular Function (MyotonPro device) (Hz) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  The Neuromuscular function will be assessed with a handheld MyotonPro myotonometry device, which will be placed on the skin, perpendicular to the surface of the belly of each gastrocnemius muscle, with the participant prone. The device will then lowered into the measurement position and held steady while it automatically conducted the predefined measurement series. The program consist of 3 single measurements with a recording interval of 1 second for each muscle. The average valuevfor each site will used in subsequent analyses. The reliability of the MyotonPro device has been reported to range from good to excellent (intraclass correlation coefficient = 0.8-0.93).
Tensomyography (m/s) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  The Tensomyography evaluation will be done by using a Dc-Dc Trans-Tek® transductor (GK 40, Panoptik d.o.o., Ljubliana, Slovenia) that will be perpendicularly placed to the gastrocnemius belly. Two self-adhesive electrodes (TMG electrodes, TMG-BMC d.o.o., Ljubljana, Slovenia) will be placed equidistant, proximal (anode) and distal (cathode) to the sensor, with an inter-electrode distance of 5 cm. Patient will be placed in prone position with a foam Electrical stimulation was applied through a TMG-100 System electrostimulator (TMG-BMCd.o.o., Ljubljana, Slovenia). The amplitude will be progressively increased from 20 to 100 mA by 20 mA increments until there will be no further increase in maximal radial displacement or maximal stimulator output was reached (i.e 110mA) (20). Ten seconds rest will be given between the stimuli to minimize the effects of fatigue and potentiation. The meters per second of muscle contraction with the electrical stimulus will be measured.

SECONDARY OUTCOMES:
Pressure Pain Threshold (Kg/cm2) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  The pressure pain threshold is the amount of pressure that is first perceived as painful. In this study, it will be assessed over the gastrocnemius TrP with a handheld mechanical pressure algometer (Trigger Plus, Pal- patronic, Hagen, Germany). Pressure will be applied at a rate of 10 N/cm2/s until the participant first reported a painful sensation. This procedure has shown good intrarater reliability.
Pain with numerical pain rating scale | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Participants will be also asked to rate their pain perception during the pressure pain threshold on an 11-point numerical pain rating scale (0 = no pain, 10 = maximum pain).
Ankle Dorsiflexion Range of Motion (º) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Active ankle dorsiflexion range of motion will be assessed with the dorsiflexion lunge test. The test will be performed by placing the foot perpendicular to a wall and lunging the knee toward the wall. The foot will be moved further away from the wall until the maximum range of dorsiflexion was achieved. In order for the heel to not lift off of the floor, the examiner will place a band under the heel and applied tension.
  The angulation from the tibia bone to the floor will be measured. The dorsiflexion lunge test has shown good intrarater and interrater reliability (intraclass correlation coefficient = 0.97).
Muscle Strentch (Newtons) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  A dynamometer (MicroFET2, Hoggan Scientific, Salt Lake City, Utah) was used for isometric muscle-strength testing. All participants will barefoot during the testing procedure. Peak force will be measured by the dynamometer to the nearest 0.1 N. Contractions will be sustained for 3 seconds while the examiner applied unmoving resistance. Both gastrocnemius-testing will be repeated for 3 trials, with a 5-second rest between them. The mean of the 3 trials will be considered in the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Pérez-Bellmunt, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No